CLINICAL TRIAL: NCT04861415
Title: A Randomized Feasibility Trial of Stereotactic Body Radiotherapy Versus Conventional Fractionation With High Dose-rate (HDR) Brachytherapy Boost for Prostate Cancer
Brief Title: SBRT vs. Conventional Fractionation With HDR Boost for Prostate Cancer
Acronym: SHARP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Gerard Morton (Other)
Responsible Party: Sponsor-Investigator, Dr. Gerard Morton, Radiation Oncologist, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2734
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Fractionated Radiation (Active Comparator): * Prostate Only Radiation - 37.5Gy in 15 daily fractions to the prostate and proximal/entire seminal vesicle
  * Prostate + Nodal Radiation - 46Gy in 23 daily fractions to the prostate, seminal vesicle and regional lymph nodes
  Interventions: Radiation: Conventionally Fractionated Radiation
- Stereotactic Body Radiotherapy (Experimental): * Prostate Only Radiation - 25Gy in 5 fractions to the prostate and proximal/entire seminal vesicle
  * Prostate + Nodal Radiation - 25Gy in 5 fractions to the prostate, seminal vesicle and regional lymph nodes
  Interventions: Radiation: Sterotactic Body Radiotherapy

INTERVENTIONS:
Radiation: Sterotactic Body Radiotherapy — Hypofractionated stereotactic radiation treatment.
  Other Names: SBRT
  Arms: Stereotactic Body Radiotherapy
Radiation: Conventionally Fractionated Radiation — External beam radiation therapy treatment
  Arms: Conventional Fractionated Radiation

SUMMARY:
Random assignment between SBRT and conventionally fractionated boost following HDR brachytherapy for prostate cancer.

DETAILED DESCRIPTION:
Many treatment options exist for prostate cancer. One common treatment approach is to combine high-dose rate (HDR) brachytherapy (temporary insertion of radiation into the prostate) and external beam radiation. External beam radiation typically requires daily radiation treatment for three to five weeks. Improvements to radiation planning and delivery has allowed stereotactic body radiation therapy (SBRT) to be implemented in many types of cancer. SBRT has been implemented as a standard treatment option after HDR brachytherapy in response to the COVID pandemic. We are seeking to evaluate whether it is feasible to randomly assign men between SBRT (which will be five treatments of radiation or conventional radiation (3-5 weeks of daily treatment) following HDR brachytherapy

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Informed consent for treatment and study participation completed
* Pathologically proven diagnosis of prostate adenocarcinoma
* ECOG Performance Status 0-2
* No prior history of pelvic radiotherapy, brachytherapy, cryosurgery, HIFU, TURP or radical prostatectomy

Exclusion Criteria:

* Presence of nodal or distant metastasis on staging MRI or CT Abdomen/Pelvis and Bone scan within 90 days of enrolment (CT/MRI/Bone Scan are only required if the clinical risk of metastatic disease is sufficient to warrant these scans)
* Plan for adjuvant chemotherapy post-radiotherapy
* Serious medical comorbidities or other contraindications to HDR brachytherapy
* Presence of inflammatory bowel disease
* Presence of connective tissue disorder seen as a contraindication to radiotherapy
* Medically unfit for general/spinal anesthesia
* Unable or unwilling to complete questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-12-23 (Actual); Primary Completion 2023-06-23 (Estimated); Study Completion 2027-12-23 (Estimated)

PRIMARY OUTCOMES:
Treatment Feasibility | 18mo - 2 years
  The proportion of patients accepting of being randomized divided by the number of patients approached for the study.

SECONDARY OUTCOMES:
QOL | 7 years
  Urinary, bowel and sexual health-related quality of life measured by the Expanded Prostate Cancer Index Composite (EPIC) domains over the study period. Each domain is normalized from 0 to 100, with a higher score indicating better outcome.
Treatment Toxicity | 7 years
  Proportion of patients with urinary, bowel and sexual Grade 2 and 3 toxicity measured by CTCAE v5.0 throughout the study period.
Cumulative biochemical failure | 7 years
  Defined as the time of enrolment to biochemical failure (based on the Phoenix definition, PSA nadir plus 2)
Overall Survival | 7 years
  Defined as time of enrollment to death from any cause
Cancer Free Survival | 7 years
  Defined as time of enrolment to death attributed to prostate cancer
Metastasis Free Survival | 7 years
  Defined as time of enrolment to development of metastasis or death from any cause
Freedom From Local Failure | 7 years
  Defined as time of enrolment to first local recurrence
Freedom From Regional Failure | 7 years
  Defined as time of enrolment to first regional recurrence
ADT Free Survival | 7 Years
  Defined as time of enrolment to salvage ADT use or death from any cause
PSA nadir | 6 years
  PSA nadir at 4-years post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Morton, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada